CLINICAL TRIAL: NCT05427097
Title: Thermal Energy of Helical® Adhesive Pads in the Treatment of Cervicogenic Dizziness
Brief Title: Thermal Energy in the Treatment of Cervicogenic Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Roseli Saraiva Moreira Bittar, Clinical Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.433.854
Record Dates: First submitted 2022-06-12; First posted 2022-06-22 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Dizziness; Cervical Pain
Keywords: Thermal; Vertigo
MeSH Terms: conditions — Dizziness; Neck Pain; Vertigo

STUDY DESIGN:
Intervention Model Description: Two groups, one placebo and one intervention
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization will be done by lottery. In a container, papers will be placed in the same number of study subjects and, then, the arm in which the subject will be allocated will be drawn. The team physiotherapist is blinded to the individual's allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): The treatment consisted of placing 10 active Helical patches spread as follows:
  * Two in the upper cervical area (suboccipital);
  * Two in the lower cervical area (near the 5th and 6th vertebrae);
  * Two in the upper trapezius muscle area (between neck and shoulder);
  * Four in the tender point area (as reported by the patient).
  Interventions: Device: Helical® patches
- Placebo (Placebo Comparator): The treatment consisted of placing 10 placebo Helical patches spread as follows:
  * Two in the upper cervical area (suboccipital);
  * Two in the lower cervical area (near the 5th and 6th vertebrae);
  * Two in the upper trapezius muscle area (between neck and shoulder);
  * Four in the tender point area (as reported by the patient).
  Interventions: Device: Helical® patches

INTERVENTIONS:
Device: Helical® patches — Active Helical® patches and non-active patches (placebo) are placed at cervical tension points
  Other Names: Non-active patches

SUMMARY:
Cervical pain contributes to postural deviations and imbalance. Nanotechnology may be used for the treatment of neck pain by fixing to the skin small rounds silicone patches containing double spiral carbon nanotubes arranged in the form of a coil (Helical), which would then relieve dizziness caused by muscular contraction.

DETAILED DESCRIPTION:
The selected patients should have neck pain arising from muscle contraction with loss of balance or instability lasting more than 90 days and normal electrooculography. Treatment consisted of placing 10 Helical patches, placebo or active, distributed as follows: two in the upper cervical area, two in the lower cervical area (near the 5th and 6th vertebrae), two in the upper trapezius muscle area (between neck and shoulder), and four in the tender point area (as reported by the patient). Using a Visual Analogue Scale (VAS) and specific questionnaires, the investigators will match pain, muscle tension and dizziness scores from Day 1 to those from Day 15 and Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Cervicogenic Dizziness diagnosis
* Normal otoneurological examination
* Signed the informed consent form
* Neck without other radiological changes, which are not solely attributable to aging (osteophytosis, rectification, disc space reduction).

Exclusion Criteria:

* Active vestibular disease
* Traumatic neck injury
* Neurological
* Rheumatic or orthopedic diseases not attributable to aging (fractures, tumors) and/or that have surgical indication
* Somatoform diseases; cognitive limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Improvement of dizziness | 60 days
  Improvement of dizziness indices provided by the visual analogue scale. Technically speaking, Visual Analog for Dizziness consists of a horizontal (or vertical) line, usually 100mm in length. The left end of the line signifies no dizziness which is depicted by a smiling face while the right end signifies the worst possible dizziness with a frowning face.

SECONDARY OUTCOMES:
Improvement of cervical neck pain | 60 days
  Improvement of cervical neck pain indices provided by the visual analogue scale.
  Technically speaking, Visual Analog for Pain consists of a horizontal (or vertical) line, usually 100mm in length. The left end of the line signifies no pain which is depicted by a smiling face while the right end signifies the worst possible pain with a frowning face.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bittar R, Alves NG, Bertoldo C, Brugnera C, Oiticica J. Efficacy of Carbon Microcoils in Relieving Cervicogenic Dizziness. Int Arch Otorhinolaryngol. 2017 Jan;21(1):4-7. doi: 10.1055/s-0036-1592418. Epub 2016 Oct 26. PMID 28050200